CLINICAL TRIAL: NCT03817827
Title: Effect of Acupuncture and Diet Modification on Amenorrhea in Female Athlete Triad
Brief Title: Effect of Acupuncture and Diet Modification on amenorrheaIN FEMALE ATHLETE TRIAD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial was delayed and patient recruitment was deemed high-risk during the Covid-19 pandemic
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Amr Hazim Abbassy, Lecturer, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 123
Record Dates: First submitted 2019-01-20; First posted 2019-01-28 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Female Athlete Triad
Keywords: sports injury; female athlete triad; acupuncture
MeSH Terms: conditions — Female Athlete Triad Syndrome; Athletic Injuries | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture (Experimental): this group will receive Acupuncture therapy for 30 minutes three times per week
  Interventions: Other: Acupuncture
- diet modification (Experimental): this group will receive diet using soy products a
  Interventions: Dietary Supplement: Diet supplementary
- combined group (Experimental): will receive both acupuncture therapy and soy products
  Interventions: Other: Acupuncture; Dietary Supplement: Diet supplementary

INTERVENTIONS:
Other: Acupuncture — this group will receive Acupuncture for 30 minutes three times per week
  Arms: Acupuncture; combined group
Dietary Supplement: Diet supplementary — Diet supplementary with soy product
  Arms: combined group; diet modification

SUMMARY:
The present study will be designed to investigate the effect of acupuncture and diet modification using soy products on amenorrhea in female athlete triad.

For this purpose this study will be carried out on sixty female athletes participating gymnastics. They will be recruited from Sports Medicine specialized center in Nasr City, their ages will range from 17 to 25 years old and their BMI will be < 20 Kg/m2 .

DETAILED DESCRIPTION:
The subjects will be divided into three groups equal in number, matched for measured variable:

Group (A): Acupuncture only will be used in this group for 30 minutes, three times per week for twelve weeks. The acupuncture needles were inserted in points located on the abdomen.

Group (B): This group will receive only the diet modification contains soy products (phytoestrogen) as 100 milliliter soy milk and 100 grams soy beans daily in the morning as a breakfast alone to ensure its absorption, this dose had been taken for 12 weeks.

Group (C): This group will receive both acupuncture therapy for 30 minutes, three times per week for 12 weeks and diet modification contains soy products as 100 milliliter soy milk and 100 grams soy beans daily in the morning for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All patients suffering from athletic amenorrhea.
* Their age will be ranged from 17-25 years old.
* Their body mass index will be less than 18.5 kg/m2.
* No history of previous pregnancies.
* No history of any pathological disease causing amenorrhea.
* They are medically stable and consented to participate in the study.

Exclusion Criteria:

* Patients with gynecological diseases that may cause amenorrhea.
* Patients using contraceptive pills.
* Patients using hormonal treatment.
* Patients using induction of ovulation methods.
* Patients following any other diet modification method.
* Patients who receive any drug with side effect of amenorrhea.

Ages: 17 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2018-05-05 (Actual); Primary Completion 2019-03-05 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
follicle stimulating hormone | three months
  Blood sample will be taken from the patient at the beginning of the study and three months later to determine the change of hormone level using Immulite 1000 immunoassay analyzer
Luteinizing hormone | three months
  Blood sample will be taken from the patient at the beginning of the study and three months later to determine the change of hormone level using Immulite 1000 immunoassay analyzer
estradiol 2 | three months
  Blood sample will be taken from the patient at the beginning of the study and three months later to determine the change of hormone level using Immulite 1000 immunoassay analyzer

CONTACTS AND LOCATIONS:
Locations (1):
- Sports medicine speciaized center, Cairo, Nasr City, Egypt